CLINICAL TRIAL: NCT03800706
Title: A Phase II Study to Evaluate the Safety and Efficacy of TQB2450 Injection in Relapsed or Refractory Classical Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2450-II-01
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Safety and Effectiveness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2450 (Experimental)
  Interventions: Drug: TQB2450

INTERVENTIONS:
Drug: TQB2450 — TQB2450 is injectived (IV) every-3-weeks (Q3W) and it should be continued until disease progression or intolerable toxicity or patients withdrawal of consent, the longest use time of experimental drugs is 96 weeks.

SUMMARY:
Single-Arm, Open-Label, Multicenter Clinical Trial. To observe the efficacy and safety of TQB2450 in patients of non-hodgkin lymphoma

ELIGIBILITY:
Inclusion Criteria:

1. Subject has voluntarily agreed to participate by giving written informed consent.;
2. Histopathological confirmed classical Hodgkin's lymphoma;
3. Relapsed/refractory cHL include：a)subject with relapse and progression after salvage chemotherapy followed by autologous stem cell transplantation(ASCT); b) subject with no ASCT: The first-line chemotherapy must be systemic multi-drug combination chemotherapy and subsequent chemotherapy requires at least one first-line chemotherapy must be systemic multi-drug combination chemotherapy; subject which is refractory didn't achieve PR after 2 cycles or didn't achieve CR after
4. Age ranged from 18 to 75 years;
5. At least one measurable disease ;
6. Patients must have ECOG performance status of 0-2;
7. Subject must have adequate organ functions ：Count of Blood Cells:hemoglobin content(HB)≥80g/L; absolute neutrophil count (ANC) ≥ 1.0 × 10^9 / L; platelet count (PLT) ≥ 75 × 10^9 / L;; Biochemical examination: serum total bilirubin (TBIL) ≤ 1.5 × normal upper limit (ULN), with the exception of patients with hepatic metastases and Gilbert's syndrome(TBIL≤3×ULN） ; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × ULN，with the exception of patients with hepatic metastases (ALT and AST ≤ 5 × ULN) , serum creatinine (Cr) ≤ 1.5 × ULN or Creatinine clearance rate（CCR）≥50 mL/min；Serum amylase and lipase ≤ 1.5 x ULN Blood coagulation function:International standardized ratio(INR)≤1.5×ULN、Activation partial thrombin time(APTT)≤1.5×ULN、Prothrombin time≤1.5×ULN；Doppler ultrasound evaluation：Left ventricular ejection fraction（LVEF)≥50%×MLN;

Exclusion Criteria:

* 1、Nodular lymphocyte-predominant Hodgkin lymphoma or gray zone lymphoma； 2、 Prior exposure to any anti-PD-1, anti-PD-L1 ， anti-CTLA-4 antibody or CAR-T cell treatment(Any other antibody that has been applied to a T cell synergistic stimulus or checkpoint pathway); 3、Need to therapy with other anticancer during the study; 4、Received allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2019-03-25 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate(ORR) | Up to 96 weeks
  Overall Response Rate (ORR) defined as the proportion of subjects who achieves a best response of CR or PR, assessed by IRC per the Lugano Classification

SECONDARY OUTCOMES:
Complete Response (CR) | Up to 96 weeks
  Disappearance of all non-target lesions and normalisation of tumour marker level. All lymph nodes must be non-pathological in size (<10mm short axis).

CONTACTS AND LOCATIONS:
Locations (1):
- No.17, panjiayuan nanli, chaoyang district, Beijing, Beijing, China